CLINICAL TRIAL: NCT01124981
Title: Efficacy and Safety of Haemocomplettan® P in Patients Experiencing Microvascular Bleeding While Undergoing Elective Complex Cardiac Surgery
Brief Title: Haemocomplettan® P During Elective Complex Cardiac Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isala (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Principal Investigator, Arno P. Nierich, MD, PhD, Isala
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BI1401_2010
Record Dates: First submitted 2010-05-10; First posted 2010-05-18 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Fibrinogen Deficiency in Complex Cardiac Surgery
Keywords: Fibrinogen concentrate; Coagulopathy
MeSH Terms: conditions — Hemostatic Disorders | interventions — Fibrinogen; Serum Albumin, Human; Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albumin (Placebo Comparator)
  Interventions: Drug: Human albumin (Placebo)
- Haemocomplettan® P (Experimental)
  Interventions: Drug: Haemocomplettan® P

INTERVENTIONS:
Drug: Haemocomplettan® P — Dosing of study medication will be individually determined based on plasma fibrinogen concentrations (measured with Clauss method during the reperfusion period on CPB) and body weight. Intravenous infusion within 10 minutes.
  Other Names: Fibrinogen concentrate
  Arms: Haemocomplettan® P
Drug: Human albumin (Placebo) — Human albumin with concentration 200g/L. The study bottles of 50 mL will be diluted with saline and will contain 2g in total. This concentration resembles the total protein load in the bottles with Haemocomplettan® P.
  Other Names: Albumin
  Arms: Albumin

SUMMARY:
Fibrinogen concentrate is increasingly used in cardiac surgery to reverse coagulopathy. Whether its use reduces blood loss, transfusion and occurrence of clinical adverse events remains unknown.

DETAILED DESCRIPTION:
Fibrinogen concentrate is increasingly used in surgical patients suffering excessive bleeding refractory to conventional hemostasis treatment. However, these studies published so far comprise small study groups with questionable study designs.

The aim of this study is to determine whether fibrinogen concentrate reduces blood loss and transfusion in patients undergoing elective complex cardiac surgery.

By choosing the domain of complex cardiac surgery which is prone for excessive blood loss and transfusion, we will focus on subjects undergoing high risk procedures. Hereby we hypothesize that administration of fibrinogen concentrate improves hemostasis in patients experiencing microvascular bleeding during complex cardiac surgery. This improvement of the hemostasis is measured by reduced blood loss and transfusion of blood products during surgery and the postoperative period.

Furthermore, we hypothesize that fibrinogen concentrate is safe and well tolerated in patients undergoing complex cardiac surgery. This hypothesis will be investigated by a detailed study of clinical outcomes.

Update regarding interim-analysis:

On 09 August 2013 an interim-analysis was performed as described in the protocol. The outcome was discussed during the Steering Committe of 09 October 2013. During that meeting, based on the results of the interim-analysis, the continuation of the current study was ordered.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older.
* Undergoing elective complex cardiac surgery.
* Understood and willingly given written informed consent.
* Experience clinically relevant non-surgical microvascular bleeding following removal of cardiopulmonary bypass.

Exclusion Criteria:

* Positive pregnancy test, pregnancy or lactation.
* Undergoing an emergency operation.
* Proof or suspicion of a congenital or acquired coagulation disorder.
* Clopidogrel use in the 5 days preceding surgery.
* INR >1.4 if on coumadin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To determine whether fibrinogen concentrate infusion reduces perioperative blood loss. | within 12 hours.
  Perioperative blood loss measured as blood loss in ml between infusion of study medication and closure of chest.

SECONDARY OUTCOMES:
To determine whether fibrinogen concentrate infusion reduces postoperative blood loss. | within 24 hours after infusion of study medication.
  Postoperative blood loss, measured as blood loss at the ICU between closure of chest and 1st hour, 6th hour and after 24 hours.
To determine whether fibrinogen concentrate infusion reduces postoperative transfusion of blood products during elective complex cardiac surgery. | within 24 hours after infusion of study medication.
  Number of units red blood cell concentrate, fresh frozen plasma and platelet concentrate administered within 24 hours after closure of chest.
To determine whether fibrinogen concentrate infusion is safe and well-tolerated. | 30 days
  Major clinical events: Mortality at 30 days post-surgery, MACE (major adverse cardiac event), cerebrovascular accident/ transient ischemic attack, renal insufficiency or failure, venous thromboembolism/ pulmonary embolism, allergic or other systemic reaction to study medication

CONTACTS AND LOCATIONS:
Overall Officials: Arno P Nierich, MD, PhD., Principal Investigator — Isala
Locations (2):
- Netherlands (2):
  - Department Anesthesiology & Intensive Care, Zwolle, Overijssel
  - Department of Cardiothoracic Anaesthesia and Intensive Care Isala Klinieken, Zwolle, Overijssel

REFERENCES:
- [Derived] Bilecen S, de Groot JA, Kalkman CJ, Spanjersberg AJ, Brandon Bravo Bruinsma GJ, Moons KG, Nierich AP. Effect of Fibrinogen Concentrate on Intraoperative Blood Loss Among Patients With Intraoperative Bleeding During High-Risk Cardiac Surgery: A Randomized Clinical Trial. JAMA. 2017 Feb 21;317(7):738-747. doi: 10.1001/jama.2016.21037. PMID 28241354
- See also: Related Info — http://www.isala.nl